CLINICAL TRIAL: NCT00060814
Title: Pilot Study Examining the Effects of Combined Pharmacotherapy (Zyban/NRT)/Behavioral Treatment on Smoking Cessation Among MMT Patients.
Brief Title: Combination Pharmacotherapy for Smoking Cessation Among Methadone Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Kimber Richter, PhD, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-00450-2; K01-00450-2
Record Dates: First submitted 2003-05-14; First posted 2003-05-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Pharmacotherapy and Counseling (Experimental): 300 mg Bupropion/4mg Nicotine Gum/Motivational Interviewing
  Interventions: Other: Combined intervention

INTERVENTIONS:
Other: Combined intervention — 300 mg bupropion plus 4mg nicotine gum ad lib plus motivational interviewing counseling

SUMMARY:
The purpose of this pilot study is to examine the effects of combined pharmacotherapy (Zyban/NRT)/behavioral treatment on smoking cessation among methadone maintenance therapy patients.

DETAILED DESCRIPTION:
This is a one-arm, open label pilot study of MMT patients to determine whether bupropion, nicotine replacement therapy, and behavioral counseling is a feasible and potentially effective intervention for smoking cessation. The smoking behaviors of participants will be be followed for 6 months post quit-date to determine effect-size estimates for a future, large scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients in long-term methadone maintenance treatment
* Patient smokes at least 10 cigarettes per day, are stable on their use of methadone (phase 2 or higher treatment), smoked for at least 1 year, be willing to participate for 6 months, and not have used bupropion or nicotine replacement therapy for 6 months

Exclusion Criteria:

* Patients who use prescription drug regimens that might affect methadone or bupropion metabolism
* Patients with cardiovascular disease, asthma, COPD
* Patients who are pregnant or breastfeeding
* Patients with regular use of alcohol, other illicit drugs, or other types of tobacco (chewing or pipe for example)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-06; Primary Completion 2002-09 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Behavioral | 6 months

SECONDARY OUTCOMES:
Number of cigarettes smoked per day | six months

CONTACTS AND LOCATIONS:
Overall Officials: Kimber Richter, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States